CLINICAL TRIAL: NCT00908752
Title: A Randomized, Double-blind, Multicenter Phase III Study of Brivanib Versus Placebo as Adjuvant Therapy to Trans-Arterial Chemo-Embolization (TACE) in Patients With Unresectable Hepatocellular Carcinoma (The BRISK TA Study)
Brief Title: Phase III Trans-Arterial Chemo-Embolization (TACE) Adjuvant HCC
Acronym: BRISK TA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA182-037; EUDRACT # 2008-008715-26
Record Dates: First submitted 2009-05-22; First posted 2009-05-27 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — brivanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brivanib (Active Comparator): Adjuvant treatment with TACE Therapy
  Interventions: Drug: Brivanib; Procedure: TACE Therapy
- Brivanib Placebo (Placebo Comparator): Placebo adjuvant treatment with TACE Therapy
  Interventions: Other: Brivanib Placebo; Procedure: TACE Therapy

INTERVENTIONS:
Drug: Brivanib — Tablets, Oral, 200 mg, once daily, until disease progression or toxicity
  Other Names: BMS-582664
  Arms: Brivanib
Other: Brivanib Placebo — Tablets, Oral, 0 mg, once daily, until disease progression or toxicity
  Arms: Brivanib Placebo
Procedure: TACE Therapy — Trans-Arterial Chemo-Embolization Therapy

SUMMARY:
The purpose of this study is to compare the Overall Survival (OS) of HCC patients who receive brivanib as adjuvant treatments to TACE therapy, with the OS of HCC patients who receive matched placebo with TACE therapy.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Patients with diagnosis of hepatocellular carcinoma
* Cirrhotic status of Child-Pugh Class A or B with a score of 7
* ECOG performance status of 0 or 1
* Adequate hematologic, hepatic, and renal function

Exclusion criteria:

* Prior use of any systemic anticancer chemotherapy, immunotherapy, investigational or molecular targeted agents for HCC
* History of cardiac disease
* Active and untreated hepatitis B
* Inability to swallow tablets or untreated malabsorption syndrome
* History of human immunodeficiency virus (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 734 (Actual)
Dates: Start 2009-07-20 (Actual); Primary Completion 2012-09-28 (Actual); Study Completion 2018-01-26 (Actual)

PRIMARY OUTCOMES:
To compare the Overall Survival (OS) of HCC patients who receive brivanib as adjuvant treatments to TACE therapy, with the OS of HCC patients who receive matched placebo with TACE therapy | Survival will be assessed continuously

SECONDARY OUTCOMES:
To compare the Time-To-Disease Progression (TTDP) of patients receiving brivanib with TACE therapy to that of patients receiving placebo with TACE therapy | Every 8 weeks
To compare the time to extrahepatic spread or vascular invasion in the brivanib and placebo arms | Every 8 weeks
To determine the total number of TACE sessions in the brivanib and placebo arms and to compare the rate of TACE sessions in the brivanib and placebo arms | End of Study
To evaluate the safety of brivanib in combination with TACE | Every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (80):
- United States (7):
  - Richard Finn, M.D., Los Angeles, California
  - Sharp Clinical Oncology Research, San Diego, California
  - Montefiore Medical Center, The Bronx, New York
  - Rhode Island Hospital, Providence, Rhode Island
  - The University Of Texas MD Anderson Cancer Center, Houston, Texas
  - University Of Virginia Health System, Charlottesville, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
- Argentina (2):
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Buenos Aires
- Local Institution, Parkville, Victoria, Australia
- Canada (2):
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Montreal, Quebec
- China (14):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Guanzhou, Guangdong
  - Local Institution, Nanning, Guangxi
  - Local Institution, Harbin, Heilongjiang
  - Local Institution, Changsha, Hunan
  - Local Institution, Changzhou, Jiangsu
  - Local Institution, Nanjing, Jiangsu
  - Local Institution, Suzhou, Jiangsu
  - Local Institution, Changchun, Jilin
  - Local Institution, Xi'an, Shan3xi
  - Local Institution, Shanghai, Shanghai Municipality
  - Local Institution, Chengdu, Sichuan
  - Local Institution, Tianjin, Tianjin Municipality
  - Local Institution, Hangzhou, Zhejiang
- France (11):
  - Local Institution, Angers
  - Local Institution, Bondy
  - Local Institution, Bordeaux
  - Local Institution, Clichy
  - Local Institution, Créteil
  - Local Institution, Grenoble
  - Local Institution, Lille
  - Local Institution, Lyon
  - Local Institution, Marseille
  - Local Institution, Paris
  - Local Institution, Toulouse
- Hong Kong (2):
  - Local Institution, Hong Kong
  - Local Institution, New Territories
- Italy (4):
  - Local Institution, Genova
  - Local Institution, Padua
  - Local Institution, Pisa
  - Local Institution, Roma
- Japan (24):
  - Local Institution, Toyoake, Aichi-ken
  - Local Institution, Chiba, Chiba
  - Local Institution, Kashiwa-shi, Chiba
  - Local Institution, Ogaki-shi, Gifu
  - Local Institution, Hiroshima, Hiroshima
  - Local Institution, Kure-shi, Hiroshima
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Kanazawa, Ishikawa-ken
  - Local Institution, Kawasaki-shi, Kanagawa
  - Local Institution, Yokohama, Kanagawa
  - Local Institution, Kochi, Kochi
  - Local Institution, Kumamoto, Kumamoto
  - Local Institution, Kyoto, Kyoto
  - Local Institution, Tsu, Mie-ken
  - Local Institution, Okayama, Okayama-ken
  - Local Institution, Higashinari-ku, Osaka
  - Local Institution, Osaka, Osaka
  - Local Institution, Ōsaka-sayama, Osaka
  - Local Institution, Sunto-gun, Shizuoka
  - Local Institution, Chuo-ku, Tokyo
  - Local Institution, Minato-ku, Tokyo
  - Local Institution, Musashino-shi, Tokyo
  - Local Institution, Toyama, Toyama
  - Local Institution, Nishinomiya-shi
- South Korea (5):
  - Local Institution, Busan
  - Local Institution, Kyunggi-do
  - Local Institution, Seoul
  - Local Institution, Suwon
  - Local Institution, Taegu
- Spain (2):
  - Local Institution, Madrid
  - Local Institution, Valencia
- Taiwan (5):
  - Local Institution, Kaohsiung City
  - Local Institution, Taichung
  - Local Institution, Tainan
  - Local Institution, Taipei
  - Local Institution, Taoyuan District
- Local Institution, Bangkok, Thailand

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm